CLINICAL TRIAL: NCT05965453
Title: Real-world Experience With the Castor Single Branch Stent Graft in the Management of Acute Aortic Syndrome
Brief Title: Evaluation of the Castor Single Branch Stent Graft in Treatment of Acute Aortic Syndrome
Acronym: ECAAS
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Hanzhong Central Hospital (Other); Affiliated Hospital of Gansu Medical College (Unknown); The Second Affiliated Hospital of Shaanxi University of Chinese Medicine (Unknown); Xianyang Hospital of Yan'an University (Unknown); Baoji Central Hospital (Other); General Hospital of Ningxia Medical University (Other); People's Hospital of Ningxia Hui Autonomous Region (Other); Qinghai Red Cross Hospital (Other); Hanzhong People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: No.XJTU1AF2023LSK-148
Record Dates: First submitted 2023-06-27; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-06

CONDITIONS: Acute Aortic Syndrome
MeSH Terms: conditions — Acute Aortic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants received thoracic endovascular aortic repair with Castor single branch stent graft: Participants who have an inadequate proximal landing zone received thoracic endovascular aortic repair by meant of the Castor single branch stent graft
  Interventions: Device: the Castor single branch stent graft

INTERVENTIONS:
Device: the Castor single branch stent graft — Participants who received thoracic endovascular aortic repair by meant of the Castor single branch stent graft from June 2018 to June 2022 were enrolled in our study.

SUMMARY:
The objective of this study to evaluate the safety and effectiveness of the Castor single branch stent graft for endovascular repair of acute aortic syndrome patients without an inadequate proximal landing zone (<15mm)

DETAILED DESCRIPTION:
The goal of this observational, ambispective, and multicenter cohort study is to evaluate efficacy and safety of the Castor single branch stent graft.

205 patients who received thoracic endovascular aortic repair by meant of the Castor single branch stent graft from June 2018 to June 2022 were enrolled in our study. All enrolled patients have an inadequate proximal landing zone (<15mm) , and they underwent routine follow-up after thoracic endovascular aortic repair at 1-month, 6-months, and 1-year for the following, but not limited to assessment: physical examination, laboratory test and the CT angiography.

Meanwhile, the enrolled patients will come for continuous follow-up at 2-years, 3-years, and annually to 10-years post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute Stanford type B aortic syndrome who received thoracic endovascular aortic repair by meant of Castor single branch stent graft from June 2018 to June 2022

Exclusion Criteria:

* Patients with acute type B aortic syndrome with an adequate proximal landing zone (≥15mm)
* Previous endovascular repair of the aorta
* Patients with missing data and loss of follow-up

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute Stanford type B aortic syndrome who received thoracic endovascular aortic repair by meant of Castor single branch stent graft in the above 10 medical centers from June 2018 to June 2022 were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 205 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2032-06-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
Immediate post-operative technique success | immediately post operation
  Immediate technical success is defined as successful delivery of the aortic and branching stent graft conveyors to their predetermined position, accurate positioning and successful deployment of the stent, safe removal of the delivery device outside the body, absence of Type I and III endoleaks on angiography at the end of the procedure, and patent branch stents.
All-cause mortality and major | 1-year post operation
  All-cause mortality includes aortic mortality, non-aortic mortality, and mortality from unknown causes.

SECONDARY OUTCOMES:
Major device/procedure-related adverse events of post-operation as assessed by computer tomography angiography | 1-month, 6-months, 1-year, and annually to 10-years post operation
  Major device or procedure related major adverse events as assessed by computer tomography angiography included: death, dissection or aneurysm rupture, new myocardial infarction requiring intervention (percutaneous transluminal coronary angioplasty, bypass), retrograde type A aortic dissection, endoleaks, new disabling stroke, paraplegia, new hepatic infarction, new chronic renal insufficiency/renal failure requiring dialysis, lower limb ischemia (increase in Rutherford classification), access vessel thrombosis or rupture, conversion to open surgery, and stent migration, fracture or migration, stent graft infection, stent graft-induced new entry tear.
Aortic remodeling results as assessed by computer tomography angiography (the size of the true and false lumen of aorta, and the thrombosis degree of the false lumen of aorta) | 1-month, 6-months, 1-year, and annually to 10-years post operation
  Compare the results of computer tomography angiography before operation and on the first-, 6th- and 12th-month post operation, the expansion of the true lumen and the thrombosis of the false lumen at the coverage of the stent graft to determine whether the blood vessel is successfully remodeled
Re-intervention during follow-up | 1-month, 6-months, 1-year, and annually to 10-years post operation
  Re-intervention result from device/procedure-related adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Tian, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No